CLINICAL TRIAL: NCT00004870
Title: A Phase I/II, Pharmacokinetic, and Biologic Correlative Study of G3139, NSC # 683428 (Phosphorothioate Antisense Oligonucleotide Directed to Bcl-2) and Irinotecan in Patients With Metastatic Colorectal Cancer
Brief Title: Olimersen and Irinotecan in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067529; SACI-IDD-98-32; UTHSC-IDD-98-32; NCI-T98-0094
Record Dates: First submitted 2000-03-07; First posted 2004-04-23 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — oblimersen; Irinotecan

INTERVENTIONS:
Biological: oblimersen sodium
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Gene therapy such as oblimersen may make tumor cells more sensitive to chemotherapy drugs. Combining irinotecan and oblimersen may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining oblimersen and irinotecan in treating patients who have metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dose-limiting toxic effects and maximum tolerated dose of augmerosen (G3139) administered in combination with irinotecan in patients with unresectable metastatic or recurrent colorectal cancer. II. Determine the quantitative and qualitative toxicity of this drug combination in this patient population. III. Assess the plasma pharmacokinetics of this combination in these patients. IV. Document the antitumor activity of this drug combination in these patients in a phase II study. V. Determine the relevant biologic endpoints of treatment in tumor biopsies prior to and after therapy with G3139 at two dose levels and assess the pharmacokinetic and pharmacodynamic correlations.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive augmerosen (G3139) IV continuously on days 1-7 and irinotecan IV over 90 minutes on day 6. Treatment continues every 21 days in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of G3139 and irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with G3139 and irinotecan at the recommended phase II dose. Patients are followed every 30 days until toxicity resolves.

PROJECTED ACCRUAL: A maximum of 18 patients will be accrued for the phase I portion of this study. A maximum of 55 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed unresectable metastatic or recurrent adenocarcinoma of the colon or rectum No brain metastases unless previously treated, asymptomatic, on stable dose of decadron, and CT/MRI scan demonstrates no evidence of edema Phase I: Measurable or evaluable disease Phase II: Measurable disease Evidence of +1 bcl-2 expression on immunohistochemical staining in pathologic material

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Absolute granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST/ALT no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases) PT/PTT normal Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection No serious concurrent systemic disorders that would preclude study treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered No other concurrent chemotherapy Phase I: At least 4 weeks since prior irinotecan and recovered Phase II: No more than 2 prior fluorouracil-based regimens for metastatic disease No prior irinotecan Endocrine therapy: See Disease Characteristics No concurrent anticancer hormonal therapy Radiotherapy: No concurrent radiotherapy Surgery: See Disease Characteristics Other: No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W. Tolcher, MD, Study Chair — San Antonio Cancer Institute
Locations (3):
- United States (3):
  - Ireland Cancer Center, Cleveland, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas